CLINICAL TRIAL: NCT06584110
Title: Effects of Buddy-Up Dyadic Physical Activity Program on Health Outcomes and Social Dynamic of Persons With Dementia and Family Caregivers: A Mixed Method Randomized Controlled Trial
Brief Title: Buddy-Up Dyadic Physical Activity Program for Persons With Dementia and Family Caregivers
Acronym: BUDPA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BUDPA-RCT
Record Dates: First submitted 2024-05-31; First posted 2024-09-04 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2024-12

CONDITIONS: Cognitive Impairment, Mild; Dementia, Mild
Keywords: dementia; dyads exercise
MeSH Terms: conditions — Cognitive Dysfunction; Dementia; Lymphoma, Follicular | interventions — Waiting Lists

STUDY DESIGN:
Intervention Model Description: BUDPA program is an overall 16-week training which comprises three phases: the conditioning, consolidating and habituating phases.
  i) Conditioning Phase (1st - 4th week) is the preparatory phase to introduce exercise movements in group training.
  ii) Consolidating Phase (5th -12th week) is the training phase for group-based exercise. Each exercise training session will be followed by a 20-minutes debriefing and goal-setting session. Self-practice will be recorded on a simple logbook.
  iii) Habituating phase (13th-16th week) aims at supporting the care dyad to integrate the partner exercises into their daily lifestyle. A video call meeting with the care dyad in week 13 and week 15 will be scheduled to offer the support.
Who Masked: Participant
Masking Description: Participants will be randomized into intervention group and wait-list control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BUDPA program (Experimental): BUDPA program is an overall 16-week training which comprises three phases: the conditioning, consolidating and habituating phases.
  i) Conditioning Phase (1st - 4th week) is the preparatory phase to introduce exercise movements in group training.
  ii) Consolidating Phase (5th -12th week) is the training phase for group-based exercise. Each exercise training session will be followed by a 20-min debriefing and goal-setting session. Self-practice will be recorded on a simple logbook.
  iii) Habituating phase (13th-16th week) aims at supporting the care dyad to integrate the partner exercises into their daily lifestyle. A video call meeting with the care dyad in week 13 and week 15 will be scheduled to offer the support.
  Interventions: Other: Buddy-Up Dyadic Physical Activity (BUDPA) program
- Usual care (Placebo Comparator): Usual care will be provided in the elderly centres. Usual care group will be put on a waiting list to receive the intervention (BUDPA program) after 24-weeks (T2) the second evaluation timepoint.
  Interventions: Other: Usual care with waiting list

INTERVENTIONS:
Other: Buddy-Up Dyadic Physical Activity (BUDPA) program — BUDPA program is an overall 16-week training which comprises three phases: the conditioning, consolidating and habituating phases.
  i) Conditioning Phase (1st - 4th week) is the preparatory phase to introduce exercise movements in group training.
  ii) Consolidating Phase (5th -12th week) is the training phase for group-based exercise. Each exercise training session will be followed by a 20-min debriefing and goal-setting session. Self-practice will be recorded on a simple logbook.
  iii) Habituating phase (13th-16th week) aims at supporting the care dyad to integrate the partner exercises into their daily lifestyle. A video call meeting with the care dyad in week 13 and week 15 will be scheduled to offer the support.
  Other Names: BUDPA
  Arms: BUDPA program
Other: Usual care with waiting list — Usual care group will be put on a waiting list to receive the intervention (BUDPA program) after 24-weeks (T2) the second evaluation timepoint.
  Arms: Usual care

SUMMARY:
The global cost of dementia is over 818 billion, and a further rise is expected in the next decade. While family caregiving is the backbone of the formal care service, promoting "living well with dementia" needs to extend to a dyadic perspective to address the needs of persons with dementia and their caregivers. Unique to dementia caregiving, imbalanced exchange in the assistance, interaction, relationship and autonomy between the partners in a care dyad always challenges their social interaction and relationships. Such eroding dyadic dynamics not only worsens the mental health of caregivers, but also compromises the quality of caregiving, fosters more dementia deterioration, and eventually complicates the caregiving process. Nevertheless, least attention is directed to dyadic dynamics in promoting living well with dementia. Partner exercise is designed in a way which requires collaboration of two members to enable the workout of each other. In addition to the benefits of exercise on dementia symptom control and caregiver's stress management, partner exercise provides a meaningful encounter to encourage reciprocity, collaboration and relationship closeness within the care dyad. This study aims to examine whether a 16-week theory-based partner exercise, named as Buddy-Up Dyadic Physical Activity (BUDPA) program, can improve dyadic dynamics and health outcomes of care dyads of mild to early-moderate dementia.

This sequential mixed-method study will recruit 111 care dyads from the elderly centers in Hong Kong. They will be randomized to receive the enhanced BUDPA program or usual care. The changes in the dyadic dynamics and health outcomes [including symptom severity and health-related quality of life (HRQL) of persons with dementia; and affect, positive aspects of caregiving and HRQL of family caregivers] between the two study groups from baseline (T0) to 16-weeks after baseline (T1) upon completion of the training , and at 24-weeks after baseline (T2). Data from outcome evaluation and interviews will be integrated to solicit a thorough understanding on the impact of BUDPA. This study marks the first attempt to use theory-driven dyadic intervention to enhance the dyadic dynamics and health outcomes of dementia care dyads. The project will advance the dyadic science in a dementia caregiving context and inform the development of evidence-based care model in dyadic fashion to promote living well with dementia in a caregiving context.

DETAILED DESCRIPTION:
The global cost of dementia is over 818 billion, and a further rise is expected in the next decade. While family caregiving is the backbone of the formal care service, promoting "living well with dementia" needs to extend to a dyadic perspective to address the needs of persons with dementia and their caregivers. Unique to dementia caregiving, imbalanced exchange in the assistance, interaction, relationship and autonomy between the partners in a care dyad always challenges their social interaction and relationships. Such eroding dyadic dynamics not only worsens the mental health of caregivers, but also compromises the quality of caregiving, fosters more dementia deterioration, and eventually complicates the caregiving process. Nevertheless, least attention is directed to dyadic dynamics in promoting living well with dementia. Partner exercise is designed in a way which requires collaboration of two members to enable the workout of each other. In addition to the benefits of exercise on dementia symptom control and caregiver's stress management, partner exercise provides a meaningful encounter to encourage reciprocity, collaboration and relationship closeness within the care dyad. This study aims to examine whether a 16-week theory-based partner exercise, named as Buddy-Up Dyadic Physical Activity (BUDPA) program, can improve dyadic dynamics and health outcomes of care dyads of mild to early-moderate dementia.

This sequential mixed-method study will recruit 112 care dyads (people with Dementia (PwD) and family caregivers) from the elderly centers in Hong Kong. They will be randomized to receive the enhanced BUDPA program or usual care.

Subject:

For people with Dementia (PwD), the inclusion criteria are i) confirmed diagnosed of dementia ii) cognitive impairment as indicated by a Hong Kong-Montreal Cognitive Assessment (Hong Kong version; HK-MoCA) score of 8-19 to indicate mild to early moderate dementia will be recruited For family caregivers, the inclusion criteria are i) live together with the PwD ii) identify as the primary family caregivers of the PwD

The changes in the dyadic dynamics and health outcomes [including symptom severity and health-related quality of life (HRQL) of persons with dementia; and affect, positive aspects of caregiving and HRQL of family caregivers] between the two study groups from baseline (T0) to 16-weeks after baseline (T1) upon completion of the training , and at 24-weeks after baseline (T2).

1. For Pwd, 4 scales will be used, Alzheimer's Disease Assessment Scale -Cognitive Subscale (ADAS-Cog), Color-Trails Test , Quality of Life-Alzheimer's Disease(QoL-AD), and The Dyadic Relationship Scale.
2. For family caregivers, measures the The Zarit Burden Interview (ZBI-C), The Neuro-psychiatric Inventory (NPI), The International Positive and Negative Affect Schedule - Short-Form (PANAS-SF 20 affect state), Medical Outcomes Study Short Form Health Survey (SF-12), The Dyadic Relationship Scale, and Positive Aspect of Caregiving Scale (PAC).

BUDPA program is an overall 16-week training which comprises three phases: the conditioning, consolidating and habituating phases.

i) Conditioning Phase (1st - 4th week) is the preparatory phase to introduce exercise movements in group training.

ii) Consolidating Phase (5th -12th week) is the training phase for group-based exercise. Each exercise training session will be followed by a 20-min debriefing and goal-setting session. Self-practice will be recorded on a simple logbook.

iii) habituating phase (13th-16th week) aims at supporting the care dyad to integrate the partner exercises into their daily lifestyle. A video call meeting with the care dyad in week 13 and week 15 will be scheduled to offer the support.

Data from outcome evaluation and interviews will be integrated to solicit a thorough understanding on the impact of BUDPA. This study marks the first attempt to use theory-driven dyadic intervention to enhance the dyadic dynamics and health outcomes of dementia care dyads. The project will advance the dyadic science in a dementia caregiving context and inform the development of evidence-based care model in dyadic fashion to promote living well with dementia in a caregiving context.

ELIGIBILITY:
Inclusion Criteria for people with dementia (PwD):

* confirmed diagnosis of dementia
* HK-MoCA score of 8-19 to indicate mild to early moderate dementia

Inclusion Criteria for family caregivers:

* live with the PwD in the same household
* self-identified as the primary family caregiver of the PwD

Exclusion Criteria for people with dementia (PwD):

* engaging in > 60 minutes per week of moderate or more vigorous exercise in the previous six months
* acute muscular-skeletal problems, stroke or cardio-respiratory disease

Inclusion Criteria for family caregivers:

* not self-identified as the primary family caregiver of the PwD

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 222 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Alzheimer's Disease Assessment Scale -Cognitive Subscale (ADAS-Cog) | baseline (T0)
  evaluate the cognitive domain function of the patient with dementia (PwD), scale from 0-70, with higher score indicating poor cognitive function.
Alzheimer's Disease Assessment Scale -Cognitive Subscale (ADAS-Cog) | 16-weeks (T1) after baseline
  evaluate the cognitive domain function of the patient with dementia (PwD), scale from 0-70, with higher score indicating poor cognitive function.
Alzheimer's Disease Assessment Scale -Cognitive Subscale (ADAS-Cog) | 24-weeks (T2) after baseline
  evaluate the cognitive domain function of the patient with dementia (PwD), scale from 0-70, with higher score indicating poor cognitive function.
Quality of Life-Alzheimer's Disease (QoL-AD) | baseline (T0)
  evaluate the health-related quality of life (HR) covering physical, functional, psychosocial, interpersonal, and environmental status of the patient with dementia, scales 13 to 52, with higher score indicating better HRQL
Quality of Life-Alzheimer's Disease (QoL-AD) | 16-weeks (T1) after baseline
  evaluate the health-related quality of life (HR) covering physical, functional, psychosocial, interpersonal, and environmental status of the patient with dementia, scales 13 to 52, with higher score indicating better HRQL
Quality of Life-Alzheimer's Disease (QoL-AD) | 24-weeks (T2) after baseline
  evaluate the health-related quality of life (HR) covering physical, functional, psychosocial, interpersonal, and environmental status of the patient with dementia, scales 13 to 52, with higher score indicating better HRQL
The Neuro-psychiatric Inventory (NPI) | baseline (T0)
  evaluate the neuro-psychiatric symptoms of the patient with dementia reported by the caregiver, scales from 12 to 96 with higher scores indicating higher severity
The Neuro-psychiatric Inventory (NPI) | 16-weeks (T1) after baseline
  evaluate the neuro-psychiatric symptoms of the patient with dementia reported by the caregiver, scales from 12 to 96 with higher scores indicating higher severity
The Neuro-psychiatric Inventory (NPI) | 24-weeks (T2) after baseline
  evaluate the neuro-psychiatric symptoms of the patient with dementia reported by the caregiver, scales from 12 to 96 with higher scores indicating higher severity
The Zarit Burden Interview (ZBI) | baseline (T0)
  evaluate the perceived caregiving burden among the caregivers, scales from 0 to 88, with higher score indicating higher perceived burden of caregivers
The Zarit Burden Interview (ZBI) | 16-weeks (T1) after baseline
  evaluate the perceived caregiving burden among the caregivers, scales from 0 to 88, with higher score indicating higher perceived burden of caregivers
The Zarit Burden Interview (ZBI) | 24-weeks (T2) after baseline
  evaluate the perceived caregiving burden among the caregivers, scales from 0 to 88, with higher score indicating higher perceived burden of caregivers
The International Positive and Negative Affect Schedule - Short-Form (PNAS-SF) | baseline (T0)
  evaluate caregiver's mood status, scales from 20 to 100, with higher score indicating higher mood change
The International Positive and Negative Affect Schedule - Short-Form (PNAS-SF) | 16-weeks (T1) after baseline
  evaluate caregiver's mood status, scales from 20 to 100, with higher score indicating higher mood change
The International Positive and Negative Affect Schedule - Short-Form (PNAS-SF) | 24-weeks (T2) after baseline
  evaluate caregiver's mood status, scales from 20 to 100, with higher score indicating higher mood change
The Color-Trails Test (CTT) | baseline (T0)
  evaluate the complex attention, executive functions and task switching for the patient with dementia, higher score indicating poor functions.
The Color-Trails Test (CTT) | 16-weeks (T1) after baseline
  evaluate the complex attention, executive functions and task switching for the patient with dementia, higher score indicating poor functions.
The Color-Trails Test (CTT) | 24-weeks (T2) after baseline
  evaluate the complex attention, executive functions and task switching for the patient with dementia, higher score indicating poor functions.
The digit span-forward and backward test | baseline (T0)
  evaluate the attention and working memory of the patient with dementia, scales from 10 to 56, with higher score indicating better attention and working memory function
The digit span-forward and backward test | 16-weeks (T1) after baseline
  evaluate the attention and working memory of the patient with dementia, scales from 10 to 56, with higher score indicating better attention and working memory function
The digit span-forward and backward test | 24-weeks (T2) after baseline
  evaluate the attention and working memory of the patient with dementia, scales from 10 to 56, with higher score indicating better attention and working memory function

SECONDARY OUTCOMES:
Medical Outcomes Study Short Form Health Survey (SF-12) | baseline (T0)
  evaluates the health-related quality of life (HRQL) of the family caregiver, scales from 12 to 60, with higher score indicating better HRQL
Medical Outcomes Study Short Form Health Survey (SF-12) | 16-weeks (T1) after baseline
  evaluates the health-related quality of life (HRQL) of the family caregiver, scales from 12 to 60, with higher score indicating better HRQL
Medical Outcomes Study Short Form Health Survey (SF-12) | 24-weeks (T2) after baseline
  evaluates the health-related quality of life (HRQL) of the family caregiver, scales from 12 to 60, with higher score indicating better HRQL
The Dyadic Relationship Scale (DRS) | baseline (T0)
  evaluate the dyadic dynamic in terms of negative relationship strain and positive interaction within the care dyad, scales from 11 to 44, with higher score indicating higher levels of dyadic strain
The Dyadic Relationship Scale (DRS) | 16-weeks (T1) after baseline
  evaluate the dyadic dynamic in terms of negative relationship strain and positive interaction within the care dyad, scales from 11 to 44, with higher score indicating higher levels of dyadic strain
The Dyadic Relationship Scale (DRS) | 24-weeks (T2) after baseline
  evaluate the dyadic dynamic in terms of negative relationship strain and positive interaction within the care dyad, scales from 11 to 44, with higher score indicating higher levels of dyadic strain
Positive Aspect of Caregiving Scale (PAC) | baseline (T0)
  evaluate caregiver's gain in terms of self -affirmation and outlook on life, scales from 0 to 44, with higher scores indicating more positive caregiving gain
Positive Aspect of Caregiving Scale (PAC) | 16-weeks (T1) after baseline
  evaluate caregiver's gain in terms of self -affirmation and outlook on life, scales from 0 to 44, with higher scores indicating more positive caregiving gain
Positive Aspect of Caregiving Scale (PAC) | 24-weeks (T2) after baseline
  evaluate caregiver&#39;s gain in terms of self -affirmation and outlook on life, scales from 0 to 44, with higher scores indicating more positive caregiving gain

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make individual participant data (IPD) available.

REFERENCES:
- [Background] Liu JD, You RH, Liu H, Chung PK. Chinese version of the international positive and negative affect schedule short form: factor structure and measurement invariance. Health Qual Life Outcomes. 2020 Aug 24;18(1):285. doi: 10.1186/s12955-020-01526-6. PMID 32838809
- [Background] Martin M, Peter-Wight M, Braun M, Hornung R, Scholz U. The 3-phase-model of dyadic adaptation to dementia: why it might sometimes be better to be worse. Eur J Ageing. 2009 Sep 29;6(4):291. doi: 10.1007/s10433-009-0129-5. eCollection 2009 Dec. PMID 28798612
- [Background] Laver K, Milte R, Dyer S, Crotty M. A Systematic Review and Meta-Analysis Comparing Carer Focused and Dyadic Multicomponent Interventions for Carers of People With Dementia. J Aging Health. 2017 Dec;29(8):1308-1349. doi: 10.1177/0898264316660414. Epub 2016 Jul 25. PMID 27458254
- [Background] Fauth E, Hess K, Piercy K, Norton M, Corcoran C, Rabins P, Lyketsos C, Tschanz J. Caregivers' relationship closeness with the person with dementia predicts both positive and negative outcomes for caregivers' physical health and psychological well-being. Aging Ment Health. 2012;16(6):699-711. doi: 10.1080/13607863.2012.678482. PMID 22548375
- [Background] Yu R, Chau PH, McGhee SM, Cheung WL, Chan KC, Cheung SH, Woo J. Trends in prevalence and mortality of dementia in elderly Hong Kong population: projections, disease burden, and implications for long-term care. Int J Alzheimers Dis. 2012;2012:406852. doi: 10.1155/2012/406852. Epub 2012 Oct 14. PMID 23097740
- [Background] Dassel KB, Carr DC. Does Dementia Caregiving Accelerate Frailty? Findings From the Health and Retirement Study. Gerontologist. 2016 Jun;56(3):444-50. doi: 10.1093/geront/gnu078. Epub 2014 Aug 26. PMID 25161263
- [Background] Stall NM, Kim SJ, Hardacre KA, Shah PS, Straus SE, Bronskill SE, Lix LM, Bell CM, Rochon PA. Association of Informal Caregiver Distress with Health Outcomes of Community-Dwelling Dementia Care Recipients: A Systematic Review. J Am Geriatr Soc. 2019 Mar;67(3):609-617. doi: 10.1111/jgs.15690. Epub 2018 Dec 10. PMID 30536383
- [Background] Law CK, Lam FM, Chung RC, Pang MY. Physical exercise attenuates cognitive decline and reduces behavioural problems in people with mild cognitive impairment and dementia: a systematic review. J Physiother. 2020 Jan;66(1):9-18. doi: 10.1016/j.jphys.2019.11.014. Epub 2019 Dec 13. PMID 31843427
- [Background] Baik D, Song J, Tark A, Coats H, Shive N, Jankowski C. Effects of Physical Activity Programs on Health Outcomes of Family Caregivers of Older Adults with Chronic Diseases: A Systematic Review. Geriatr Nurs. 2021 Sep-Oct;42(5):1056-1069. doi: 10.1016/j.gerinurse.2021.06.018. Epub 2021 Jul 11. PMID 34261027
- [Background] Yu HM, He RL, Ai YM, Liang RF, Zhou LY. Reliability and validity of the quality of life-Alzheimer disease Chinese version. J Geriatr Psychiatry Neurol. 2013 Dec;26(4):230-6. doi: 10.1177/0891988713500586. Epub 2013 Aug 22. PMID 23970459
- [Background] Leung VP, Lam LC, Chiu HF, Cummings JL, Chen QL. Validation study of the Chinese version of the neuropsychiatric inventory (CNPI). Int J Geriatr Psychiatry. 2001 Aug;16(8):789-93. doi: 10.1002/gps.427. PMID 11536346
- [Background] Ko KT, Yip PK, Liu SI, Huang CR. Chinese version of the Zarit caregiver Burden Interview: a validation study. Am J Geriatr Psychiatry. 2008 Jun;16(6):513-8. doi: 10.1097/JGP.0b013e318167ae5b. PMID 18515696
- [Background] Moyle W, Jones C, Dwan T, Ownsworth T, Sung B. Using telepresence for social connection: views of older people with dementia, families, and health professionals from a mixed methods pilot study. Aging Ment Health. 2019 Dec;23(12):1643-1650. doi: 10.1080/13607863.2018.1509297. Epub 2018 Nov 17. PMID 30450924
- [Background] Lam CL, Tse EY, Gandek B. Is the standard SF-12 health survey valid and equivalent for a Chinese population? Qual Life Res. 2005 Mar;14(2):539-47. doi: 10.1007/s11136-004-0704-3. PMID 15892443
- [Background] Sebern MD, Whitlatch CJ. Dyadic relationship scale: a measure of the impact of the provision and receipt of family care. Gerontologist. 2007 Dec;47(6):741-51. doi: 10.1093/geront/47.6.741. PMID 18192628
- [Background] Lou VW, Lau BH, Cheung KS. Positive aspects of caregiving (PAC): scale validation among Chinese dementia caregivers (CG). Arch Gerontol Geriatr. 2015 Mar-Apr;60(2):299-306. doi: 10.1016/j.archger.2014.10.019. Epub 2014 Nov 7. PMID 25488014
- [Background] Vallejo G, Fernandez MP, Livacic-Rojas PE, Tuero-Herrero E. Selecting the best unbalanced repeated measures model. Behav Res Methods. 2011 Mar;43(1):18-36. doi: 10.3758/s13428-010-0040-1. PMID 21287107
- [Background] Elo S, Kyngas H. The qualitative content analysis process. J Adv Nurs. 2008 Apr;62(1):107-15. doi: 10.1111/j.1365-2648.2007.04569.x. PMID 18352969
- [Background] Wolf ZR. Exploring the audit trail for qualitative investigations. Nurse Educ. 2003 Jul-Aug;28(4):175-8. doi: 10.1097/00006223-200307000-00008. PMID 12878896
- [Background] Younas A, Pedersen M, Durante A. Characteristics of joint displays illustrating data integration in mixed-methods nursing studies. J Adv Nurs. 2020 Feb;76(2):676-686. doi: 10.1111/jan.14264. Epub 2019 Nov 25. PMID 31713252